

Reshaping the future of patient care

November 10, 2022

Martha Kruhm, MS RAC Head, Protocol and Information Office Quality Assurance Section CTEP, DCT, NCI 6130 Executive Blvd, EPN Room 7000 Bethesda, MD 20892

Dear Ms. Kruhm:

Enclosed is Addendum #31 to EAY131-V, MATCH Treatment Subprotocol V: Phase II Study of Sunitinib in Patients with Tumors with cKIT Mutations (Excluding GIST, Renal Cell Carcinoma or Pancreatic Neuroendocrine Tumor).

Please replace your current copy of the protocol and Informed Consent document with these updated versions. We recommend that each institution maintain a file containing the original protocol, Informed Consent, and all subsequent revisions/versions.

#### **IRB Review Requirements:**

This addendum has been reviewed and approved by the Central IRB, which is the sole IRB of record for this study. Local IRB review and approval is unnecessary.

**Implementation of this addendum must occur on the activation date.** Sites are not permitted to conduct the study utilizing outdated versions of any MATCH protocol documents after the activation date of this addendum.

The following revisions to the EAY131-V protocol have been made in this addendum:

| | Section | Change |
|---|---|---|
| 1. | Cover Page | Updated Version Date and addendum number. |
| 2. | Contact<br>Page | Updated the phone number for the subprotocol chair, Dr. Lilian Gien. |

The following revisions to the EAY131-V Informed Consent Document have been made in this addendum:

| | Section | Change |
|----|------------|-----------------------|
| 1. | Cover Page | Updated Version Date. |

If you have any questions regarding this addendum, please contact <u>eradomyshelsky@ecogacrin.org</u> or 857-504-2900.

| We request review and approval of this addendum to EAY131-V so ECOG-ACRIN may activate it promptly. |
|---|
| Thank you. |
| Sincerely, |
| Pamela Cogliano |

Senior Director of Protocol Development

# Study Title for Study Participants: Testing Sunitinib as potentially targeted treatment in cancers with cKIT genetic changes

## Official Study Title for Internet Search on http://www.ClinicalTrials.gov/:

Molecular Analysis for Therapy Choice (MATCH)

MATCH Treatment Subprotocol V: EAY131-V: Phase II Study of Sunitinib in Patients with Tumors with c-Kit Mutations (Excluding GIST, Renal Cell Carcinoma or Pancreatic Neuroendocrine Tumor).

Version Date: November 10, 2022

#### Rev. Add25 What is the usual approach to my cancer?

You are being asked to take part in this part of the study because you have genetic changes in your tumor that are potentially targeted by Sunitinib. There is currently no agreed upon approach for treating cancers with the genetic changes, called either a cKIT, a PDGFR- $\alpha$ , or a PDGFR- $\beta$  mutation that you have. People who are not in a study are usually treated with either surgery, radiation, or with drugs that have been FDA approved. Sometimes, combinations of these are used and your doctor can explain which may be best for you. These treatments can reduce symptoms and may stop the tumor from growing for several months or more.

## What are my other choices if I do not take part in this study?

If you decide not to take part in this study, you have other choices. For example:

- you may choose to have the usual approach described above
- you may choose to take part in a different study, if one is available
- or, you may choose not to be treated for cancer but you may want to receive comfort care to relieve symptoms

Version Date: November 10, 2022

## Rev. Add25 Why is this study being done?

The purpose of this study is to test any good and bad effects of the study drug, Sunitinib, in patients whose cancer has genetic changes called cKIT, PDGFR- $\alpha$ , or PDGFR- $\beta$  mutations. Sunitinib could shrink your cancer, but it could also cause side effects. Researchers hope to learn if Sunitinib will shrink the cancer by at least one-quarter compared to its present size. Sunitinib has been approved by the FDA for use in renal cell (kidney) cancer, pancreatic neuroendocrine tumor and for gastrointestinal stromal tumors (GIST). The use of Sunitinib for the treatment of other cancers with cKIT, PDGFR- $\alpha$ , or PDGFR- $\beta$  mutations is considered experimental. There will be about 35 people taking part in this study.

Rev. 2/16 Rev. 3/17

## What are the study groups?

All study participants will get the same study drug, Sunitinib. Sunitinib should be taken for 4 weeks continuously, regardless of ideal or actual body weight, followed by 2 weeks of rest. Swallow capsules whole. Do not crush, chew or open capsules. If you forget to take your scheduled dose, the missed pills will not be taken later.

You will be required to maintain a patient pill calendar and bring it with you to every clinic visit.

A study calendar that shows how often exams, tests, and/or procedures will be done is attached

## How long will I be in this study?

You will receive the study drug as long as your cancer does not get worse, the side effects are tolerable and you agree to stay on study. When you finish taking Sunitinib, your doctor will continue to watch you for side effects and follow your condition with visits to the office for follow-up exams every 3 months for 2 years and then every 6 months for the third year from your enrollment in the study.

## What possible risks can I expect from taking part in this study?

If you choose to take part in this study, there is a risk that:

- You may lose time at work or home and spend more time in the hospital or doctor's office than usual
- You may be asked sensitive or private questions which you normally do not discuss

Sunitinib used in this study may affect how different parts of your body work such as your liver, kidneys, heart, thyroid and blood. The study doctor will be testing your blood and will let you know if changes occur that may affect your health. These risks are described in more detail below.

There is also a risk that you could have other side effects from the study drug.

Here are important points about side effects:

• The study doctors do not know who will or will not have side effects.

- Some side effects may go away soon, some may last a long time, or some may never go away.
- Some side effects may interfere with your ability to have children.
- Some side effects may be serious and may even result in death.

Here are important points about how you and the study doctor can make side effects less of a problem:

- Tell the study doctor if you notice or feel anything different so they can see if you are having a side effect.
- The study doctor may be able to treat some side effects.
- The study doctor may adjust the study drugs to try to reduce side effects.

The tables below show the most common and the most serious side effects that researchers know about. There might be other side effects that researchers do not yet know about. If important new side effects are found, the study doctor will discuss these with you.

Rev. 5/16 Rev. 3/17 Rev. Add21

#### Possible Side Effects of Sunitinib malate

(Table Version Date: February 15, 2019)

#### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving sunitinib malate (SU011248 L-malate), more than 20 and up to 100 may have:

- Pain
- Constipation, diarrhea, heartburn, nausea, vomiting
- Sores in the mouth
- Tiredness
- Loss of appetite
- Changes in taste
- Sore throat
- Redness, pain or peeling of palms and soles

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving sunitinib malate (SU011248 L-malate), from 4 to 20 may have:

- Anemia which may require blood transfusion
- Blurred vision with chance of blindness
- Bloating, passing gas
- Dry mouth, skin
- Chills, fever
- Swelling of arms, legs
- Flu-like symptoms including body aches
- Bruising, bleeding

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving sunitinib malate (SU011248 L-malate), from 4 to 20 may have:

- Weight loss
- Infection, especially when white blood cell count is low
- Dehydration
- Dizziness, headache
- Feeling of "pins and needles" in arms and legs
- Depression
- Difficulty sleeping
- Cough, shortness of breath
- Nose bleed
- Hair loss, rash, itching, skin changes
- Change in hair color
- High blood pressure which may cause headaches, dizziness, blurred vision

#### RARE, AND SERIOUS

In 100 people receiving sunitinib malate (SU011248 L-malate), 3 or fewer may have:

- Anemia, kidney problems which may cause tiredness, bruising, swelling, or may require dialysis
- Blood clot which may cause confusion, paralysis, seizures or swelling, pain, shortness of breath
- Damage to organs (heart, brain, others) which may cause shortness of breath, swelling of ankles, and tiredness, changes in thinking
- Heart failure, heart attack which may cause shortness of breath, swelling of ankles, and tiredness
- Pain and swelling of thyroid
- Visual loss
- Difficulty swallowing
- A tear or hole in or between internal organs which may cause drainage and may require surgery
- Swelling of the gallbladder
- Liver damage which may cause yellowing of eyes and skin, swelling
- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Flesh-eating bacteria syndrome
- Non-healing surgical site
- Change in the heart rhythm
- Kidney damage which may require dialysis
- Damage to the jawbone which may cause loss of teeth

- Damage to muscle which may cause muscle pain, dark red urine
- Cancer of bone marrow caused by chemotherapy
- Damage to the bone marrow (irreversible) which may cause infection, bleeding, may require transfusions
- Stroke
- Brain damage which may cause headache, seizure, blindness (also known as Reversible Posterior Leukoencephalopathy Syndrome)
- Sores on the skin
- Severe skin rash with blisters and peeling which can involve mouth and other parts of the body

Let your study doctor know of any questions you have about possible side effects. You can ask the study doctor questions about side effects at any time.

You should report and discuss with the study doctor any other medication(s) you are taking while you are treated with the study drugs, so that he/she can take action to prevent any potential drug interactions.

Please refer to the drug interaction handout and wallet card for additional information.

#### Rev. 3/17 **Reproductive risks:**

You should not become pregnant, breastfeed, or father a baby while in this study. The drugs in this study could be very damaging to an unborn baby. Check with the study doctor about what types of birth control, or pregnancy prevention, to use while in this study.

It is important that you understand that you need to either practice "abstinence" (that is avoiding sexual activity) or use birth control while on this study.

Avoiding sexual activity is the only certain method to prevent pregnancy. However, if you choose to be sexually active, you must agree to use an appropriate double barrier method of birth control (such as female use of a diaphragm, intrauterine device (IUD), sponge and spermicide, in addition to the male use of a condom) or involve female use of prescribed "birth control pills" or a prescribed birth control implant. Both double barrier contraception and birth control pills or implants must be used for at least one week prior to the start of the study and continuing for 16 weeks after the last dose of the study drugs. If you choose to be sexually active during the study, you must accept that pregnancy could still result, exposing you or your sexual partner to potential loss of pregnancy as well as other unknown effects on the developing unborn baby. If a woman becomes pregnant while on this study or within 4 weeks after the last dose of study drug, she will be asked for information concerning the outcome of her pregnancy. If a female partner of a male patient becomes pregnant while the male patient is on the study or within 4 weeks after the last dose of study drug, the male patient must notify the investigator.

## What possible benefits can I expect from taking part in this study?

This study has only a small chance of helping you because we do not know if the study drug/study approach is effective. This study may help researchers learn things that may help other people in the future.

## Can I stop taking part in this study?

Yes. You can decide to stop at any time. If you decide to stop for any reason, it is important to let the study doctor know as soon as possible so you can stop safely. If you stop, you can decide whether or not to let the study doctor continue to provide your medical information to the organization running the study.

The study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

The study doctor may take you out of the study:

- If your health changes and the study is no longer in your best interest
- If new information becomes available such that it is in your interest to stop investigational treatment
- If you do not follow the study rules
- If the study is stopped by the sponsor, IRB or FDA.

## If your cancer becomes worse during treatment with the study drug:

- You may be asked to take part in another MATCH study treatment. Your study doctor will discuss this with you.
- Another biopsy may be required and will be tested to determine if your tumor has new genetic changes and if there is another MATCH study treatment available for your cancer as described in the MATCH Screening Consent.
- This testing will be similar to the testing for genetic changes that was done in the initial screening step of this study.
- Your study doctor will be given the results of these new genetic tests and share them with you.
- There may be some additional exams or procedures required for this next treatment. These will be discussed in a separate Consent Form about the next treatment that you will receive.

## What are my rights in this study?

Taking part in this study is your choice. No matter what decision you make, and even if your decision changes, there will be no penalty to you. You will not lose medical care or any legal rights.

## What are the costs of taking part in this study?

**ECOG-ACRIN** 

The Sunitinib will be supplied at no charge while you take part in this study. It is possible that the Sunitinib may not continue to be supplied while you are on the study. Although not likely, if this occurs, your study doctor will talk to you about your options.

You and/or your health plan/insurance company will need to pay for all of the other costs of treating your cancer while in this study, including the cost of study drug preparation and administration (if any), and tests, procedures, or medicines to manage any side effects, unless you are told that certain tests are being done at no charge. Before you decide to be in the study, you should check with your health plan or insurance company to find out exactly what they will pay for.

You will not be paid for taking part in this study.

## What happens if I am injured or hurt because I took part in this study?

If you are injured or hurt as a result of taking part in this study and need medical treatment, please tell your study doctor. The study sponsors will not offer to pay for medical treatment for injury. Your insurance company may not be willing to pay for study-related injury. If you have no insurance, you would be responsible for any costs.

If you feel this injury was a result of medical error, you keep all your legal rights to receive payment for this even though you are in a study.

## Who will see my medical information?

Your privacy is very important to us and the researchers will make every effort to protect it. Your information may be given out if required by law. For example, certain states require doctors to report to health boards if they find a disease like tuberculosis. However, the researchers will do their best to make sure that any information that is released will not identify you. Some of your health information, and/or information about your specimen, from this study will be kept in a central database for research. Your name or contact information will not be put in the database.

The ECOG-ACRIN Cancer Research Group is carrying out this study. ECOG-ACRIN is a cancer research group that conducts studies for the National Cancer Institute. Your doctor is a member of ECOG-ACRIN or another group that is participating in this study. To help protect your privacy, ECOG-ACRIN has obtained a Confidentiality Certificate from the U.S. Department of Health and Human Services (DHHS). With this Certificate, ECOG-ACRIN cannot be forced (for example, by court subpoena) to disclose information that may identify you in any federal, state or local civil, criminal, administrative, legislative or other proceeding. Disclosure will be necessary, however, upon request of DHHS for audit or program evaluation purposes.

There are organizations that may inspect your records. These organizations are required to make sure your information is kept private, unless required by law to provide information. Some of these organizations are:

The study sponsor and the drug company supporting the study.

- The Institutional Review Board, IRB, is a group of people who review the research with the goal of protecting the people who take part in the study.
- The Food and Drug Administration and the National Cancer Institute in the U.S., and similar ones if other countries are involved in the study.

## Where can I get more information?

Date of signature

You may visit the NCI Web site at <a href="http://cancer.gov/">http://cancer.gov/</a> for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

| Who | o can answer my questions about | t this study? | |
|---|---|---|---|
| | You can talk to the study doctor about any preport side effects or injuries. Contact of study doctor[s]) at | | |
| My | signature agreeing to take part i | n the main study | |
| a | have read this consent form or had it reand my questions have been answered. I wake part in the main study. | | • |
| P | articipant's signature | | |
| _ | | | |
| Γ | Date of signature | | |
| S | ignature of person(s) conducting the infe | ormed consent discussion | |

Rev.2/16 Rev. 3/17

## **Study Calendar**

| Visit | Patient Activities |
|---|---|
| Before starting study drugs (within four to six weeks of start of treatment) | <ul> <li>Routine blood tests</li> <li>Urine tests</li> <li>Electrocardiogram (ECG)</li> <li>Echocardiogram (ECHO) or nuclear study (Multigated Acquisition [MUGA] or similar scan) to assess your heart function, if clinically necessary</li> <li>Pregnancy test (if you are a woman who could become pregnant)</li> <li>History and physical examination</li> <li>Imaging (CT or MRI; same method to be used at future visits)</li> </ul> |
| Week 1:<br>Day 1 | <ul> <li>History and physical examination, if they have not been completed within 7 days</li> <li>Routine blood tests, if they have not been completed within 7 days</li> <li>Urine tests, if they have not been completed within 7 days</li> <li>Begin taking Sunitinib, the study drug</li> </ul> |
| Week 2:<br>Day 8 | Blood pressure measurements |
| Week 3:<br>Day 15 | Blood pressure measurements |
| Week 3:<br>Day 21 (± 3 days) | <ul><li>History and physical examination</li><li>Routine blood tests</li><li>Urine tests</li></ul> |
| Week 6<br>Day 36 | Blood pressure measurements |
| Week 7:<br>Day 1 | <ul> <li>History and physical examination</li> <li>Routine blood tests</li> <li>Urine tests</li> <li>Electrocardiogram (ECG), if clinically necessary</li> <li>Return pills and patient pill calendar</li> </ul> |
| Week 9:<br>Day 21 (± 3 days) | <ul> <li>History and physical examination</li> <li>Routine blood tests</li> <li>Urine tests</li> </ul> |

**EAY131-V** 

| Week 13 (and onwards): | • Every 6 weeks: Routine blood tests, a history of how you feel, a physical examination, an ECG (if clinically necessary), and urine tests |
|---|---|
| Day 1 | • Every 12 weeks (while you are on the study): Imaging (CT or MRI; by same method as screening) |
| | • Every 12 weeks (while you are on the study): Echocardiogram (ECHO) or nuclear study (Multigated Acquisition [MUGA] or similar scan) to assess your heart function, if clinically necessary |
| | Every 6 weeks: Return pills and patient pill calendar at each clinic visit |
| End of treatment | Side effects assessment |
| | Return pills and patient pill calendar |
| Follow up: | History and physical examination |
| Every three months | Side effects assessment, if clinically necessary |
| for two years and | Routine blood tests, if clinically necessary |
| every six month for<br>the third year | <ul> <li>Imaging (CT or MRI; by same method as screening), if clinically<br/>necessary</li> </ul> |